CLINICAL TRIAL: NCT05085652
Title: Is SARS-CoV-2 (Covid-19) a Risk Factor for Hypotension During Spinal Anesthesia for Obstetric Patients?
Brief Title: Spinal Anesthesia Related Hypotension in SARS-CoV-2 (COVID-19) Pregnant Patients
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Aygun cuhadar, anesthesiology and reanimation specialist, MD, primer investigator, Ankara City Hospital Bilkent
Other Study IDs: 72300690-799-1
Record Dates: First submitted 2021-10-10; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hypotension; Regional Anesthesia Morbidity; SARS-CoV2 Infection
Keywords: spinal anesthesia; regional anesthesia for SARS-CoV-2; spinal anesthesia induced hypotension
MeSH Terms: conditions — Hypotension; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypotensive COVID19 patients: Neuraxial anesthesia-related hypotension was based on a single episode of deﬁned hypotension from the time of local anesthetic injection until 15 min after delivery of the newborn. And hypotension was deﬁned as systolic blood pressure <80% of baseline or <90 mmHg and was treated with an intravenous bolus of ephedrine 5 mg, additional bolus of Ringer Lactates and colloid infusion hydroxyethyl starch solution.
  Interventions: Procedure: spinal anesthesia induced hypotension in SARS-CoV-2 patients.
- non-hypotensive COVID19 patients: from the time of local anesthetic injection until 15 min after delivery of the newborn no hypotension was seen. systolic blood pressure > 80% of baseline or >90 mmHg. no medical treatment needed.

INTERVENTIONS:
Procedure: spinal anesthesia induced hypotension in SARS-CoV-2 patients. — SARS-CoV-2 infection prognosis remains unclear during pregnancy. according to ESA, ASRA and WHO regional anesthesia was recommended to use for caesarian section procedures. But at the beginning of the pandemic Chen et al shared their retrospective analyses about regional anesthesia for caesarian section and they showed high spinal anesthesia induced hypotension in 14 patients of the 17 and also again Chen and Zahng et al made another study and this time they found 57,4% hypotension incidence. In our study we aimed to find if the spinal anesthesia safe procedure in the 249 patients and one center hospital.
  Groups: hypotensive COVID19 patients

SUMMARY:
Since the onset of COVID-19, recommendations suggest the use of neuraxial anesthesia, if possible, over general anesthesia for cesarian section to avoid the risks of aerosolization associated with tracheal intubation and extubation. But the safety of performing spinal anesthesia is unclear especially for post spinal hypotension, during the presence of active infection with COVID-19. Since at the beginning of the pandemic a few studies reported significant hypotension during epidural anesthesia in COVID-19 pregnant women, there was a controversial discussion about the safety of regional anesthesia was started. In this study we aimed to find if spinal anesthesia is safely recommended anesthesia type for COVID-19 obstetric patients. 249 patients with PCR confirmed COVID-19 for cesarean section undergoing spinal anesthesia in Ankara City Hospital, Ankara assessed in this retrospective study to find if the hypotension is the risk factor for the COVID-19 patients.

DETAILED DESCRIPTION:
The emergence of severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2) which defined coronavirus disease 2019 (COVID-19) has prompted innumerable alterations in practice of anesthesiology. The nature of the association between COVID-19 and pregnancy outcomes remains unclear, and meta-analyses involving patients with COVID-19 who are pregnant are limited. A 2020 systematic review suggested that people who are pregnant did not have an increased risk of SARS-CoV-2 infection or symptomatic COVID19, but they were at risk of severe COVID-19 compared with those who were not. But unlike previous viral pandemics, COVID-19 incidence, prognosis and maternal and neonatal outcomes do not appear to be worse in pregnant women compared to that general population.

All of the potential complications of COVID 19 for pregnant and especially higher rate of aerosol transmission to the healthcare persons The American Society of Regional Anesthesia --- ASRA, the European Society of Regional Anesthesia and Pain Medicine --- ESRA and the European Society of Anesthesiology ---ESA published guidance on employing regional anesthesia for patients with COVID-19.

With regional anesthesia the risk of person-to-person transmission, which is 6,6 times higher during the respiratory procedures performed in general anesthesia getting minimalized.

In cesarean section for pregnant women with COVID-19 infection, all the questions for if the spinal anesthesia was safe and efficient in achieving satisfactory obstetrical anaesthesia? At the beginning of the pandemic in a retrospective analysis Chen et al reported that higher rate of hypotension after neuraxial blocks. After this study some questions about safety of the regional anesthesia appeared in the minds.

However, the eﬀects of SARS-CoV-2 infection on hemodynamics of pregnancies who underwent neuraxial anesthesia for cesarean delivery are still unclear. In this study we retrospectively evaluated 249 COVID-19 patients in one center hospital in case the hypotension is the risk for the neuraxial block safety and if so, what we did to treat them?

Method:

After the approval of the local ethical committee approval, we used a retrospective analysis of 249 COVID 19 cesarean section spinal anesthesia to determine the incidence of hypotension and management strategies after the anesthesia. The study was carried out with the principles of the Helsinki Declaration. Medical records of pregnant women who were admitted into our hospital for cesarean section were retrospectively retrieved during the period of January 24, 2020 - February 29, 2021. The diagnosis criteria followed the guideline by the National Health Commission of Turkey and SARS-CoV-2 nucleic acid test was used to screen COVID-19 in all patients. All ASA Physical Status II pregnant women who received cesarean delivery under neuraxial anesthesia were eligible for inclusion in the study.

Neuraxial anesthesia protocols for cesarean delivery was before the spinal anesthesia, an intravenous line, ECG, pulse oximetry, and non-invasive automatic blood pressure monitors (2-min interval) were placed. Spinal anesthesia was performed in the sitting position with 26-gauge atraucan spinal needle and heavy bupivacaine regards of the anesthesiologists through the L3-4 or L4-5 intervertebral spaces. All patients were delivered oxygen by nasal cannula under the surgical mask. All the patients placed in the supine position after puncture procedure until the end of the surgical procedure. All BP recordings in this study were performed with the patient in the supine position.

Neuraxial anesthesia-related hypotension was based on a single episode of deﬁned hypotension from the time of local anesthetic injection until 15 min after delivery of the newborn. And hypotension was deﬁned as systolic BP <80% of baseline or <90 mmHg and was treated with an intravenous bolus of ephedrine 5 mg, additional bolus of Ringer Lactates and colloid infusion hydroxyethyl starch solution (130/0.46% hydroxyethyl starch solution; Fresenius Kabi, Bad Homburg vor der Höhe, Germany). All the demographic-vital data's including systolic and diastolic blood pressure (SBP-DBP), ephedrine-atropine doses, crystalloids and colloid infusion volumes, newborn birth weight and nausea, vomiting was recorded too.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 nucleic acid test positive COVID-19 all ASA Physical Status I- II pregnant women who received cesarean delivery under neuraxial anesthesia were eligible for inclusion in the study.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: SARS-CoV-2 nuclec acid test positive ASA I-II pregnant who scheduled to cesarian section operations.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
hypotension | From the time of local anesthetic injection to subarachnoid space until 15 min after delivery of the newborn.
  Systolic Blood Pressure <80% of baseline or <90 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Aygün Güler, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Aygün Güler, Ankara, Type A Choice Below ..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Clinical Study Report — https://doi.org/10.1007/s12630-020-01630-7 — Chen R, Zhang Y, Huang L, Cheng B, Xia Z, Meng Q. Safety and efﬁcacy of different anesthetic regimens for parturients with COVID-19 undergoing cesarean delivery: a case series of 17 patients. Can J Anesth. 2020. DOI: https://doi.org/10.1007/s12630-020-01630-7
- Available data/document: Clinical Study Report — https://dx.doi.org/10.3389%2Ffmed.2021.713733 — 12- Zhang Y, Chen R, Cao C, et al. The Risk of Neuraxial Anesthesia-Related Hypotension in COVID-19 Parturients Undergoing Cesarean Delivery: A Multicenter, Retrospective, Propensity Score Matched Cohort Study. Front Med (Lausanne). 2021;8:713733. Published 2021 Aug 19. doi:10.3389/fmed.2021.713733